CLINICAL TRIAL: NCT01710514
Title: A Multi-Center, Randomized, Open-Label, Parallel Group Study of FE 999913 Vaginal Tablet 100 mg in Japanese Female Patients Undergoing Fertility Treatment [In Vitro Fertilization/Embryo Transfer (IVF-ET)]
Brief Title: A Phase III Study of FE 999913 in Japanese Female Patients Undergoing Fertility Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000072
Record Dates: First submitted 2012-10-09; First posted 2012-10-19 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Luteal Hormone Supplementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FE 999913 100 mg BID (Active Comparator): FE 999913 100 mg vaginal tablet BID
  Interventions: Drug: FE 999913 vaginal tablet
- FE 999913 100 mg TID (Active Comparator): FE 999913 100 mg vaginal tablet TID
  Interventions: Drug: FE 999913 vaginal tablet

INTERVENTIONS:
Drug: FE 999913 vaginal tablet

SUMMARY:
The purposes of the study are to verify sufficient supplementation of luteal hormone after administrating FE999913 Vaginal Tablet twice a day (BID) or three times a day (TID) and to determine the efficacy and safety of FE999913 Vaginal Tablet in Japanese women undergoing fertility treatment with IVF-ET (a fresh embryo transfer).

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal adult women between the ages of 20 and 42 years.
* Early follicular phase (day 2-4) follicle stimulating hormone (FSH) ≤12 IU/L and Estradiol <100 pg/mL.
* Luteinizing hormone (LH), prolactin (PRL), and thyroid-stimulating hormone (TSH), within the normal limits for the clinical laboratory tests, or considered not clinically significant by the investigator within 6 months prior to screening.
* Documented history of infertility [e.g., unable to conceive for at least one year (or for 6 months for women ≥38 years of age) or bilateral tubal occlusion or absence].
* Transvaginal ultrasound at screening (or within 14 days prior to screening) consistent with findings adequate for Assisted Reproduction Technology (ART) with respect to uterus and adnexa (peripheral reproductive organs).
* At least one cycle with no fertility medication prior to screening.
* Hysterosalpingography, hysteroscopy, sonohysterogram, or transvaginal ultrasound documenting a normal uterine cavity.
* Consent to contraception during the cycle in which pituitary down regulation is performed (prior to start of controlled ovarian stimulation).
* Signed informed consent to fertility treatment using FE999913 Vaginal Tablet after the subject and her husband have thoroughly understood the content.

Exclusion Criteria:

* Donor oocyte or embryo recipient; gestational or surrogate carrier.
* Undergoing blastomer biopsy and other experimental ART procedures.
* Severe hepatic dysfunction or disease.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Porphyria.
* Presence of any clinically relevant systemic disease (eg, insulin-dependent diabetes mellitus).
* Past or current surgical or medical condition which in the judgment of the Principal Investigator (or Sub-investigator) may interfere with absorption, distribution, metabolism, or excretion of the study drug.
* Subjects with a body mass index (BMI) of >34 at time of Screening.
* Previous IVF or ART failure due to a poor response to gonadotropins*.

  * Defined as development of ≤2 mature follicles or history of 2 previous cycle cancellations prior to oocyte retrieval due to poor response.
* Presence of abnormal uterine bleeding of undetermined origin.
* Current or recent (within the past 12 months) substance abuse, including alcohol.
* Known or suspected breast or genital tract cancer.
* History of chemotherapy or radiotherapy for malignant disorder (chorionic disease).
* Currently breast feeding, pregnant or contraindication to pregnancy.
* Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled visits and clinical laboratory tests.
* Documented intolerance or allergy to any of the medications to be used in the study including the investigational medicinal product.
* Participation in any experimental drug study within 60 days prior to Screening.
* Use of any of the following medications during the pretreatment and treatment phase: hormonal drug products (use of oral contraceptives prior to start of controlled ovarian stimulation is allowed), other progesterone drug products, hydrocortisone and other steroid drug products, and fertility modifiers such as insulin sensitizers.
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (6):
- Japan (6):
  - Hanabusa Women's Clinic, Kobe, Hyōgo
  - Ebina Ladies Clinic, Ebina, Kanagawa
  - Sophia Ladies Clinic, Sagamihara, Kanagawa
  - Bashamichi Ladies Clinic, Yokohama, Kanagawa
  - IVF Namba Clinic, Osaka, Osaka
  - Sanno Hospital, Tokyo

REFERENCES:
- [Derived] Fujiwara T. A multi-center, randomized, open-label, parallel group study of a natural micronized progesterone vaginal tablet as a luteal support agent in Japanese women undergoing assisted reproductive technology. Reprod Med Biol. 2015;14(4):185-193. doi: 10.1007/s12522-015-0211-y. Epub 2015 Jun 14. PMID 26457065

RESULTS

PARTICIPANT FLOW:
Groups:
- FE 999913 100 mg BID: FE 999913 100 mg vaginal tablet BID
  FE 999913 vaginal tablet
- FE 999913 100 mg TID: FE 999913 100 mg vaginal tablet TID
  FE 999913 vaginal tablet
Period: Overall Study
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID
Started | 54 | 54
Intent-To-Treat (ITT) Analysis Set | 54 (All randomised subjects were included in the Intent-To-Treat (ITT) analysis set.) | 54 (All randomised subjects were included in the ITT analysis set.)
Full Analysis Set (FAS) | 46 (All randomised and exposed subjects with at least one completed primary efficacy assessment.) | 48 (All randomised and exposed subjects with at least one completed primary efficacy assessment.)
FAS With Embryo Transfer (ET) | 43 (Data on pregnancy was reported for the subjects with embryo transfer.) | 47 (Data on pregnancy was reported for the subjects with embryo transfer.)
Safety Analysis Set | 54 (All subjects received at least one dose of Investigational Medicinal Product (IMP).) | 54 (All subjects received at least one dose of IMP.)
Completed | 47 | 47
Not Completed | 7 | 7
Not completed — Adverse Event | 6 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population
Groups:
- Total: Total of all reporting groups
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] — FAS population
  years | 34.9 (3.6) | 34.5 (4.25) | 34.7 (3.93)
Age, Customized [Number; unit: participants] — FAS population
  participants
    <35 years | 17 | 21 | 38
    35-37 years | 17 | 14 | 31
    38-40 years | 11 | 8 | 19
    41-42 years | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — FAS population
  Participants
    Female | 46 | 48 | 94
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 46 | 48 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Day of transfer [Number; unit: participants] — FAS with embryo transfer (ET) (BID: 43, TID: 47, Total: 90)
  participants
    Day 3 | 38 | 45 | 83
    Day 5 | 5 | 2 | 7
Subjects with embryo transferred [Number; unit: participants] — FAS with ET (BID: 43, TID: 47, Total: 90)
  participants
    1 embryo | 39 | 42 | 81
    2 embryos | 4 | 5 | 9
Embryos transferred [Mean (Standard Deviation); unit: embryos] — FAS with ET (BID: 43, TID: 47, Total: 90)
  embryos | 1.09 (0.294) | 1.11 (0.312) | 1.1 (0.302)
Method of insemination [Number; unit: participants] — FAS with ET (BID: 43, TID: 47, Total: 90)
  participants
    IVF | 19 | 21 | 40
    Intracytoplasmic Sperm Injection (ICSI) | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Blood Progesterone Concentration Not Less Than 10 ng/ml
Time Frame: Day 5 of treatment
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- FE999913 000072 (BID/TID): Data pooled from both BID and TID groups
Arm/Group | FE999913 000072 (BID/TID)
Number analyzed (Participants) | 94
percentage of subjects | 98.9 [94.2 to 100.0]
Statistical Analysis 1: Comparison: FE999913 000072 (BID/TID); To verify sufficient supplementation of luteal hormone, the proportion of subjects with blood progesterone concentration ≥ 10 ng/mL on Day 5 was compared to the result from a historical control, trial CS08 (NCT number: 00884221). The corresponding proportion of subjects in trial CS08 was 99.8% (95%CI: 99.1;100.0, 631/632 subjects). The non-inferiority hypothesis tested for this primary endpoint was: H0: P(000072)-P(CS08) ≤ -10.0% against the alternative Ha: P(000072)-P(CS08) > -10.0%; Test type: Non-Inferiority or Equivalence — The null hypothesis (H0) was tested against the alternative (Ha) by constructing two-sided 95%CI for the difference. The non-inferiority limit for the difference was pre-specified to -10.0% (absolute). If the lower limit of the two-sided 95%CI was greater than the non-inferiority limit (-10.0%) for both the FAS and per protocol set, the null hypothesis was to be rejected. In that case it would be claimed that the rate observed in this trial was non-inferior to the rate observed in the CS08 trial; Difference of % to historical control = -0.9, 95% CI 2-sided [-3.6 to 1.8]

2. Primary Outcome: Ongoing Pregnancy Rate
Description: Defined as identification of fetal survival and fetal heart movements on transvaginal ultrasound
Time Frame: Week 5 of study
Population: FAS with ET population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FE 999913 Total: Data pooled from BID and TID groups
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | FE 999913 Total
Number analyzed (Participants) | 43 | 47 | 90
percentage of participants | 14.0 [5.3 to 27.9] | 29.8 [17.3 to 44.9] | 22.2 [14.1 to 32.2]

3. Secondary Outcome: Rate of Positive βeta Human Chorionic Gonadotrophin (βhCG)
Time Frame: Week 2 of study
Population: FAS with ET population In the TID group 13 subjects had a positive beta-hCG assessment while 14 subjects had a positive clinical pregnancy at Week 4. This is because one subject had a negative beta-hCG at Week 2, but she had a positive local serum hCG on the same day and continued the trial. Then clinical and ongoing pregnancy were confirmed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | FE 999913 Total
Number analyzed (Participants) | 43 | 47 | 90
percentage of participants | 16.3 [6.8 to 30.7] | 27.7 [15.6 to 42.6] | 22.2 [14.1 to 32.2]

4. Secondary Outcome: Clinical Pregnancy Rate
Description: Defined as presence of a gestational sac on transvaginal ultrasound
Time Frame: Week 4 of study
Population: FAS with ET population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | FE 999913 Total
Number analyzed (Participants) | 43 | 47 | 90
percentage of participants | 14.0 [5.3 to 27.9] | 29.8 [17.3 to 44.9] | 22.2 [14.1 to 32.2]

5. Secondary Outcome: Blood Progesterone Concentration
Time Frame: Weeks 2, 4, 5, 8, and end of study
Population: FAS population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | FE 999913 Total
Number analyzed (Participants) | 46 | 48 | 94
ng/mL
  Baseline; n=46, 48, 94 | 0.626 (0.379) | 0.704 (0.364) | 0.666 (0.371)
  Week 2; n=32, 42,74 | 11.4 (12.0) | 30.7 (37.9) | 22.3 (31.0)
  Week 4; n=6, 14, 20 | 32.5 (23.1) | 77.9 (41.3) | 64.2 (42.0)
  Week 5; n=6, 14,20 | 32.3 (17.0) | 67.7 (35.7) | 57.1 (35.0)
  Week 8; n=5, 12, 17 | 41.4 (15.7) | 53.3 (23.5) | 49.8 (21.7)
  End of study; n=38, 46, 84 | 10.8 (16.3) | 21.9 (26.4) | 16.9 (23.0)

ADVERSE EVENTS:
Arm/Group | FE 999913 100 mg BID | FE 999913 100 mg TID | FE 999913 Total
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/54 | 1/108
Other Adverse Events (participants affected / at risk) | 15/54 | 22/54 | 37/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999913 100 mg BID (N=54) | FE 999913 100 mg TID (N=54) | FE 999913 Total (N=108)
Subchorionic haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999913 100 mg BID (N=54) | FE 999913 100 mg TID (N=54) | FE 999913 Total (N=108)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 2 (4)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 10 (10) | 12 (12) | 22 (22)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.